CLINICAL TRIAL: NCT06907186
Title: A Single-arm Interventional Pilot Study to Investigate the Feasibility and Acceptance of a Structured Psychological Support Program for Patients, Caregivers, and Presymptomatic Carriers in Hereditary Transthyretin Amyloidosis With Cardiomyopathy
Brief Title: An Interventional Pilot Study to Investigate the Feasibility and Acceptance of a Structured Psychological Support Program for Patients, Caregivers, and Presymptomatic Carriers in Hereditary Transthyretin Amyloidosis With Cardiomyopathy
Acronym: AMH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Laura Obici, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AMH
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Transthyretin Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Hereditary Transthyretin Amyloidosis (Other): Patient with Hereditary Transthyretin Amyloidosis
  Interventions: Other: Psychological Support

INTERVENTIONS:
Other: Psychological Support — Carrying out a systematic and organized path of psychological support interviews on a monthly basis in person or remotely.

SUMMARY:
Hereditary transthyretin amyloidosis (ATTRv) is a genetic, progressive and disabling disease that affects multiple organs and severely compromises the quality of life of patients and their families. A holistic approach is essential, which, in addition to early diagnosis and clinical management, includes psychological support to address the emotional and psychosocial impact of the disease. Although specific interventions for mental well-being are recommended, studies evaluating support tools for patients with ATTRv cardiomyopathy and their caregivers are lacking.

DETAILED DESCRIPTION:
The overall objective of the study is to evaluate the feasibility, acceptance and preliminary efficacy data of a structured psychological support program for patients, caregivers and presymptomatic carriers in hereditary transthyretin amyloidosis (ATTRv) with cardiomyopathy.

The primary objective is to evaluate the feasibility of a psychological support program for patients, caregivers and presymptomatic carriers.

The co-primary objective is to evaluate the acceptance by patients of the proposed psychological support program.Key secondary objective: Evaluate the effects of the psychological support program on the levels of anxiety and depression in patients and presymptomatic carriers of ATTRv during the psychological support pathway (at 6 months) and at the end (at 12 months);

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years;
* Fluent in Italian;
* Patient, presymptomatic carrier or ATTRv caregiver, in charge of UOC General Medicine 2 - Amyloidosis Center of the Fondazione IRCCS Policlinico San Matteo in Pavia;
* Signing of the specific Informed Consent

Exclusion Criteria:

* Subjects who, although belonging to UOC General Medicine 2 - Amyloidosis Center of the Fondazione IRCCS Policlinico San Matteo in Pavia - present a diagnosis of another type of amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The feasibility of a psychological support program | 12 months
  measured by calculating the percentage of interviews in which the patient participates, at least 80%.
Acceptance of a psychological support program | 12 months
  Acceptability will be assessed based on how many T0 patients accept psychological support

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Medicina Generale 2 - Centro Amiloidosi Sistemiche e Malattie ad Alta Complessità, Pavia, Italy